CLINICAL TRIAL: NCT05430841
Title: Evaluating the Potential Usefulness of 18F-AlF-FAPI PET/CT in Patients With Gastrointestinal Tumors and Compared With 18F-FDG PET/CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XMYY-2021KY061
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer; Pancreatic Cancer; Liver Cancer
Keywords: Diagnosis; Positron-Emission Tomography; Gastric Cancer; Pancreatic Cancer; Liver Cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-AlF-FAPI PET/CT (Experimental): Each subject receives a single intravenous injection of 18F-FDG and 18F-AlF-FAPI, and undergo PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: 18F-FDG, 18F-AlF-FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG, 18F-AlF-FAPI PET/CT — Each subject receives a single intravenous injection of 18F-FDG and 18F-AlF-FAPI, and undergo PET/CT imaging within the specified time.

SUMMARY:
To evaluate the potential usefulness of 18F-AlF-FAPI positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in gastrointestinal tumors, and compared with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Subjects with gastrointestinal tumors underwent contemporaneous 18F-AlF-FAPI and 18F-FDG PET/CT either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The numbers of positive tumor lesions of 18F-FDG and 18F-AlF-FAPI PET/CT were recorded by visual interpretation. The sensitivity, specificity, and accuracy of 18F-AlF-FAPI, 18F-FDG PET/CT were calculated and compared to evaluate the diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years or order);
* patients with suspected or newly diagnosed or previously treated gastrointestinal tumors (supporting evidence may include MRI, CT, tumor markers and pathology report);
* patients who had scheduled both 18F-FDG and 18F-AlF-FAPI PET/CT scans;
* patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* patients with non-malignant lesions;
* patients with pregnancy;
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 30 days
  The sensitivity, specificity, and accuracy of 18F-FDG and 18F-AlF-FAPI PET/CT were calculated and compared to evaluate the diagnostic efficacy.

SECONDARY OUTCOMES:
SUV | 7 days
  Standardized uptake value (SUV) of 18F-FDG and 18F-AlF-FAPI PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.
Number of lesions | 7 days
  The numbers of positive primary and metastatic lesions of 18F-FDG and 18F-AlF-FAPI PET/CT were recorded by visual interpretation.

CONTACTS AND LOCATIONS:
Overall Officials: Long Sun, PhD, Study Chair — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First affiliated hospital of xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu W, Cai J, Peng T, Meng T, Pang Y, Sun L, Wu H, Zhang J, Chen X, Chen H. Fibroblast Activation Protein-Targeted PET/CT with 18F-Fibroblast Activation Protein Inhibitor-74 for Evaluation of Gastrointestinal Cancer: Comparison with 18F-FDG PET/CT. J Nucl Med. 2024 Jan 2;65(1):40-51. doi: 10.2967/jnumed.123.266329. PMID 37884330